CLINICAL TRIAL: NCT05470803
Title: An Observer-blind, Cohort Randomized, Exploratory Phase 3 Study to Evaluate the Safety and Immunogenicity of Recombinant Covid-19 Vaccine (AstraZeneca/Fiocruz), mRNA Covid-19 (Comirnaty, Pfizer/Wyeth) Vaccine and Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2019-Clover) as 4th Dose in Individuals Primed/ Boosted With Various Regimens
Brief Title: An Observer-blind, Cohort Randomized, Exploratory Phase 3 Study to Evaluate the Safety and Immunogenicity of Recombinant Covid-19 Vaccine, mRNA Covid-19 Vaccine and Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine as 4th Dose in Individuals Primed/ Boosted With Various Regimens
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TP-SCB-2019-002
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a phase 3, cohort randomized, observer-blind, multi-center study to evaluate the safety and immunogenicity of a 4th dose of the following SARS-CoV-2 vaccines: recombinant COVID-19 vaccine -AstraZeneca/Fiocruz, mRNA covid-19 vaccine - Pfizer/Wyeth and SCB-2019-Clover.
Who Masked: Participant
Masking Description: This study will be observer-blind. Due to the visual differences between the SCB-2019/Clover, Recombinant Covid-19 (AstraZeneca/Fiocruz) and mRNA Covid-19 (Comirnaty, Pfizer/Wyeth) study vaccines, the participants will be blinded before receiving the study vaccination. An unblinded dosing team, not involved with study participant's evaluation, will prepare and administer the study vaccines.
  The investigational product syringe will be opacified to avoid unblinding of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A: 03 doses Pfizer/Wyeth (Experimental): Group 1: AstraZeneca/Fiocruz Group 2: Pfizer/Wyeth Group 3: Clover SCB-2019
  Interventions: Biological: AstraZeneca/Fiocruz; Biological: Pfizer/Wyeth; Biological: Clover SCB-2019
- Cohort B: 03 doses AstraZeneca/Fiocruz (Experimental): Group 4: AstraZeneca/Fiocruz Group 5: Pfizer/Wyeth Group 6: Clover SCB-2019
  Interventions: Biological: AstraZeneca/Fiocruz; Biological: Pfizer/Wyeth; Biological: Clover SCB-2019
- Cohort C: 03 doses Sinovac/Butantan or 02 doses and 01 dose AstraZeneca/Fiocruz (Experimental): Group 7: AstraZeneca/Fiocruz Group 8: Pfizer/Wyeth Group 9: Clover SCB-2019
  Interventions: Biological: AstraZeneca/Fiocruz; Biological: Pfizer/Wyeth; Biological: Clover SCB-2019
- Cohort D: 02 doses AstraZeneca/Fiocruz and 01 dose Alum/CpG adjuvanted 9 or 30 µg Clover SCB-2019 (Experimental): Group 10: Clover SCB-2019
  Interventions: Biological: Clover SCB-2019

INTERVENTIONS:
Biological: AstraZeneca/Fiocruz — 4th dose of SARS-CoV-2 vaccine
  Arms: Cohort A: 03 doses Pfizer/Wyeth; Cohort B: 03 doses AstraZeneca/Fiocruz; Cohort C: 03 doses Sinovac/Butantan or 02 doses and 01 dose AstraZeneca/Fiocruz
Biological: Pfizer/Wyeth — 4th dose of SARS-CoV-2 vaccine
  Arms: Cohort A: 03 doses Pfizer/Wyeth; Cohort B: 03 doses AstraZeneca/Fiocruz; Cohort C: 03 doses Sinovac/Butantan or 02 doses and 01 dose AstraZeneca/Fiocruz
Biological: Clover SCB-2019 — 4th dose of SARS-CoV-2 vaccine

SUMMARY:
This is an exploratory phase 3, cohort randomized, observer-blind, multi-center study to evaluate the safety and immunogenicity of a 4th dose of various SARS-CoV-2 vaccines. There will be 04 study cohorts, that have previously received 03 doses of the indicated vaccine (s), divided into 10 groups; and each one of the 10 study groups will receive the 4th dose. This exploratory study will enroll up to 360 participants in 4 cohorts and a total of 10 groups: Cohort A (N=90), Cohort B (N= 90), Cohort C (N=150) and Cohort D (N=30). In cohorts A-C participants will be randomized 1:1:1 to three different 4th dose regimens. The number of proposed participants will provide a reasonable accurate descriptive summary of the safety and immunogenicity of the tested vaccination regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age. Participation of individuals >60 years will be limited to ≤ 10/ group.
2. Individuals are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests, and other study procedures.
3. Individuals are willing and able to give an informed consent, prior to screening.

   * Individuals who received one of the following vaccination regimens 3 doses of Pfizer/ Wyeth; 3 doses of AstraZeneca/Fiocruz; or 2 doses of Sinovac/Butantan and 1 dose of AstraZeneca, or eventually 3 doses of Sinovac/Butantan; or 2 doses of AstraZeneca and 1 dose of Alum/CpG-adjuvanted 9 µg or 30 µg Clover SCB-2019 vaccine (participants of study TP-SCB-2019-002).
   * Interval between last priming dose and 3rd dose minimum 3 months
   * Interval between 3rd dose and 4th dose ≥ 4 months
4. Healthy participants or participants with pre-existing medical conditions who are in a stable medical condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
5. Female participants are eligible to participate in the study if not pregnant, not breastfeeding, and at least 1 of the following criteria apply:

   * Women of non-childbearing potential;
   * Women of childbearing potential (WOCBP) must have a negative urine pregnancy test prior to study vaccination. A confirmatory serum pregnancy test may be conducted at the investigator's discretion. They must be using a highly effective licensed method of birth control for 30 days prior to the first vaccination and must agree to continue such precautions during the study until 90 days after the last study vaccination.
6. Male participants must agree to employ acceptable contraception from the day of dose of the study vaccine until 6 months after the last dose of the study vaccine/comparator and also refrain from donating sperm during this period.

Exclusion Criteria:

1. Individuals with fever >37.5°C (axillary), or any acute illness at baseline (Day 0) or within 3 days prior to randomization. Participants meeting this criterion may be rescheduled within the relevant window. Febrile participants with minor illnesses can be enrolled at the discretion of the investigator.
2. Individuals who have received more than 3 combined doses of any licensed or experimental COVID vaccine prior to Day 0 or plan to receive COVID-19 vaccine during the study period, a drug for COVID-19 prevention or treatment (e.g., drugs, monoclonal antibodies, such as Rituximab or any other anti-CD20 monoclonal antibodies during the study period.).
3. Receipt of any authorized or investigational COVID-19 vaccine prior to Day 0 except for the 03 doses of Pfizer/ Wyeth; 03 doses of AstraZeneca/Fiocruz; or two doses of Sinovac/Butantan and 01 dose of Pfizer/Wyeth, or eventually 03 doses of Sinovac/Butantan; or two doses of AstraZeneca and one dose of Clover SCB-2019 ≥ 4 months before enrollment in this study.
4. Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction (e.g., anaphylaxis) to any component of the study vaccines (Pfizer/Wyeth, AstraZeneca/Fiocruz, CpG 1018, aluminum, or SCB-2019 components as outlined in the latest summary of product characteristics for Pfizer/Wyeth, AstraZeneca/Fiocruz and the IB for SCB-2019.
5. Individuals with known bleeding disorder that would, in the opinion of the investigator, contraindicate intramuscular injection.
6. Individuals who have a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix which have been cured, or other malignancies with minimal risk of recurrence).
7. Individuals with any progressive or severe neurologic disorder, seizure disorder, or history of Guillain-Barré syndrome.
8. Individuals who received treatment with immunosuppressive therapy in the last 90 days, including cytotoxic agents or systemic corticosteroids, or planned receipt during the study period. If a short-term course of systemic corticosteroid immunosuppressive dose has been used for the treatment of acute illness, the participant should not be included in the study until corticosteroid therapy has been discontinued for at least 15 days prior to first study vaccination. If the participant has used an immunosuppressive dose of a depot corticosteroid, intra-muscular or intra-articular, they must wait 60 days for inclusion in the study. Inhaled or nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
9. Individuals with autoimmune diseases, except: Hashimoto's thyroiditis, vitiligo, psoriasis, lupus discord and alike; HIV-positive individuals and/or on HIV treatment.
10. Individuals who have received any other investigational product within 30 days prior to Day 0 or intend to participate in another clinical study at any time during the conduct of this study.
11. Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 28 days after the last vaccination.
12. Individuals who have received treatment with Rituximab or any other anti-CD20 monoclonal antibodies within 9 months prior to Day 0 or planned during the study period.
13. Administration of intravenous immunoglobulins and/or any blood products within 3 months prior to enrollment or planned administration during the study period.
14. Individuals with any condition that, in the opinion of the investigator, would interfere with the primary study objectives or pose additional risk to the participant.
15. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | 28 days after the administration of a 4th dose of anti-COVID-19 vaccines
  VNA positivity and Anti-Spike IgG antibody titers (ELISA) for several strains of SARS-CoV2 (Wuhan, Delta, Omicron BA.1, optionally BA.4/5 and/or BA.1.12) at baseline (day 0) and day 28 after 4th dose.

SECONDARY OUTCOMES:
Immunogenicity | 84 days after the administration of a 4th dose of anti-COVID-19 vaccines
  VNA positivity and Anti-Spike IgG antibody titers (ELISA) for several strains of SARS-CoV-2 (Wuhan, Delta, Omicron BA.1, optionally BA.4/5 and/or BA.1.12) at baseline (day 0) and day 84 after 4th dose.

OTHER OUTCOMES:
Safety: Occurrence of SAEs, AESIs and severe unsolicited AEs | At days 28 and 84
  Occurrence of SAEs, AESIs and severe unsolicited AEs
Safety: Total and severe local / systemic solicited AEs | At days 0 to 7
  Total and severe local / systemic solicited AEs
Number of SARS-CoV-2 infection cases | At days 28 and 84
  Occurrence of confirmed episodes of COVID-19 by RT-PCR or lateral flow test

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Centro de Estudos e Pesquisa em Moléstias Infecciosas (CEPCLIN), Natal, Rio Grande do Norte
  - Crie Unifesp, São Paulo, São Paulo
  - Hospital Gloria D'or, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Undecided